CLINICAL TRIAL: NCT04000737
Title: A Phase II Randomized Placebo-Controlled Study Investigating The Combination Of YIV-906 And Sorafenib (Nexavar®) In HBV (+) Patients With Advanced Hepatocellular Carcinoma
Brief Title: YIV-906 (Formerly PHY906/KD018) With Sorafenib in HBV(+) Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yiviva Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YIV-906-2018L1
Record Dates: First submitted 2019-06-13; First posted 2019-06-27 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Advanced Adult Hepatocellular Carcinoma; BCLC Stage B Adult Hepatocellular Carcinoma; BCLC Stage C Adult Hepatocellular Carcinoma; Hepatitis B (+) Associated Advanced Hepatocellular Carcinoma; Child-Plough A Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B | interventions — PHY 906

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sorafenib + YIV-906 (Experimental): Patients in the study arm will be treated orally for 28-day courses with YIV-906 + sorafenib
  Interventions: Drug: Sorafenib+YIV-906
- Sorafenib + Placebo (Active Comparator): Patients in the placebo arm will be given sorafenib with placebo
  Interventions: Drug: Sorafenib+placebo

INTERVENTIONS:
Drug: Sorafenib+YIV-906 — Patients will be given sorafenib (400 mg BID) daily for a 28-day course with YIV-906 (3 capsules, BID) 4 days on and 3 days off weekly in each course.
  Other Names: PHY906; KD018
  Arms: Sorafenib + YIV-906
Drug: Sorafenib+placebo — Patients will be given sorafenib (400 mg BID) daily for a 28-day course with placebo (3 capsules, BID) 4 days on and 3 days off weekly in each course.
  Arms: Sorafenib + Placebo

SUMMARY:
The aim of this study is to compare the efficacy and safety of YIV-906 plus standard-of-care sorafenib versus those of sorafenib alone as a first-line systemic treatment for patients with Hepatitis B (+) associated advanced hepatocellular carcinoma.

YIV-906 (PHY906, KD018) is an immune system modulator. Clinical and preclinical research suggests that YIV-906 could act to enhance the body's immune response to fight cancer and increase the anti-tumor activity of sorafenib and protect and repair the gastrointestinal tract by reducing inflammation and promoting tissue regeneration.

Inspired by a 1,800-year-old traditional medicine still in use today, YIV-906 is a botanical drug candidate, composed of an extract of four herbs and administered in oral capsule form.

The CALM (Combination of YIV-906 and Sorafenib to treat Advanced Liver cancer in a Multi-center study) trial is a multi-regional, randomized, placebo-controlled study.

DETAILED DESCRIPTION:
HCC patients with chronic HBV (+) (HBsAg(+)), and Child-Pugh A status will be randomized to either the study arm (YIV-906 plus sorafenib) or control arm (placebo plus sorafenib) at ratio of 2:1. Patients will be stratified according to metastatic status (extrahepatic/vascular invasion vs. none), and their ECOG performance status (0 vs. 1) at randomization.

* ARM I: Patients receive Placebo + Sorafenib
* ARM II: Patients receive YIV-906+ Sorafenib

Patients in the study arm will be treated orally each 28-day course with YIV-906 (600 mg (3 capsules) BID) + sorafenib (400 mg BID) according to the following schedule: sorafenib BID daily treatment for 28 days, and YIV-906 BID 4 days on and 3 days off weekly in each course.

All patients will be evaluated and graded for adverse events according to the NCI Common Terminology for Adverse Events, version 5.0 (CTCAE). The Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) will be used to establish disease response or progression.

The RECIST 1.1 and mRECIST will be used in a blinded independent central review (BICR) to determine the study endpoints.

Patients will be evaluated for PFS, TTP, OS, antitumor response every two cycles, and QoL and safety at the beginning of each cycle. Biomarkers are mandatory and will be studied prior to drug administration on day 1 of each cycle. TCM Syndrome Research is optional.

PK is only applicable in China study sites and limited to the first 15 male and 15 female patients. Patients will be randomized to either the study drug arm or the placebo arm (2:1 ratio). PK studied immediately prior to dose administration and at 1 hour, 2 hours, 4 hours, and 12 hours post-dose administration on Day 1 of Cycles 1.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females ≥18 years old with ability to take oral drugs
2. Diagnosis of advanced (locally advanced or metastatic) unresectable/inoperable HCC according to the American Association for the Study of Liver Diseases (AASLD) Guidelines (Heimbach et al. 2018) or diagnosis by tissue pathology
3. Participants categorized to stage B or C based on Barcelona Clinic Liver Cancer (BCLC) staging system
4. Life expectancy of at least 3 months
5. Presence of chronic hepatitis B (HBsAg (+))
6. Never received systemic antitumor therapy
7. Patients must have at least one tumor lesion that meets both of the following criteria:

   1. "Measurable disease" according to RECIST1.1, i.e. at least one measurable lesion.
   2. Advanced unresectable HCC that have liver limited disease who have failed and are not candidates to local therapies; or patients with extrahepatic disease.
8. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
9. Cirrhotic status of current Child-Pugh class A. Child-Pugh status should be calculated based on clinical findings and laboratory results during the screening period
10. For patients with positive HBV-DNA and positive HBsAg, they must be treated with anti-HBV treatment (per local standard of care), as prophylaxis starting at least 1-2 weeks prior to receiving study drug and willing to continue treatment for the length of the study
11. Patients with adequate organ reserve, such as laboratory parameters:

    1. Absolute Neutrophil Count (ANC) ≥ 1.5 x 10^9/L
    2. Platelets ≥ 60000 x 10^6/L
    3. Hemoglobin (Hgb) ≥ 9 g/dL
    4. Serum alanine amino-transferase (ALT) ≤ 5 x ULN
    5. Serum Aspartate transaminase (AST) ≤ 5 x ULN
12. Adequate renal function, based upon meeting the following laboratory criteria within 7 days before randomization:

    1. Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 40mL/min (using the Cockcroft-Gault equation: (140-age) x weight (kg)/ (serum creatinine x 72 [mg/dL] for males. (For females multiply by 0.85) AND
    2. Urine protein/creatine ratio (UPCR) ≤ 1 mg/mg (≤113.1 mg/mmol) or 24-hour urine protein <1 g
13. Ability to understand and willingness to sign a written informed consent and to be able to follow the visit schedule

Exclusion Criteria:

Patient who has any of the following criteria will be excluded from the trial:

1. Patients who ever have HCV infection
2. Patients who have received systemic chemotherapies or immunotherapy or molecular target therapies or anticancer Chinese medicine Cinobufacini
3. Patients who have received any local anti-cancer therapy within 4 weeks prior to Cycle 1 treatment
4. Active bleeding (including gastrointestinal bleeding) during the last 4 weeks prior to Cycle 1 treatment
5. Patients with a history of allergy to the known components of YIV-906
6. Known history of human immunodeficiency virus (HIV) seropositivity
7. Known central nervous system metastasis including brain metastasis and meningeal carcinomatosis
8. Hepatocholangiocarcinoma, fibrolamellar cell carcinoma and mixed hepatocellular carcinoma
9. Active malignancy (except for definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma-in-situ of the cervix) within the past 5 years
10. Any severe and/or uncontrolled medical conditions including but not limiting:

    1. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤ 6 months prior to Cycle 1 treatment, serious uncontrolled cardiac arrhythmia, uncontrolled hypertension
    2. Previous transient ischemic attack (TIA), cerebral vascular accident (CVA), symptomatic peripheral vascular disease (PVD) within last 6 months of Cycle 1 treatment
    3. Congenital long QT syndrome
    4. Alcoholic patients
    5. Acute and chronic, active infectious disorders and nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy, in the opinion of the investigator, except chronic HBV
    6. Impairment of gastrointestinal function or who have gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
    7. Patients who have had organ transplantation
11. Patients receiving chronic treatment with corticosteroids (except for intermittent topical or local injection of aldosterone) or other immunosuppressive agents (oral prednisone or equivalent 10 mg/day is allowed to screen).
12. Patients received any blood transfusion, albumin transfusion, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF), TPO or other medical supportive treatment within 4 weeks of Cycle 1 treatment
13. Patients treated with drugs known to be strong inducers of isoenzyme CYP3A within 7 days of Cycle 1 treatment
14. Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from surgery
15. Patients who have received an investigative drug or therapy within the last 4 weeks prior to Cycle 1 treatment
16. Pregnant and/or breastfeeding women
17. Men and women of childbearing age and potential, who are not willing to use effective contraception
18. Unwilling or unable to follow protocol requirements or to give informed consent
19. Ongoing or recent history of autoimmune, uncontrolled psychiatric disorders and drug abuse
20. Uncontrolled hereditary or acquired thrombotic or bleeding disorder
21. Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection
22. Therapeutic dose anticoagulation with warfarin, or similar agents
23. Chronic therapy with nonsteroidal anti-inflammatory agents or other anti-platelet agents. Aspirin at doses up to 100 milligrams/day is permitted
24. No patient, however, may enroll in this trial if they are taking phenytoin (Dilantin)
25. Patients taking traditional Chinese medicines within 14 days prior to taking first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | At baseline, then at the end of every two cycle (i.e. approximately every 8 weeks), until disease progression or discontinuation from study. Assessed up to 24 months.
  PFS is defined as the period elapsing between the date of date of randomization and the date of either disease progression or date of death, whichever is earlier.

SECONDARY OUTCOMES:
Time to progression (TTP) | At baseline, then at the end of every two cycle (i.e. approximately every 8 weeks), until disease progression or discontinuation from study. Assessed up to 24 months.
  TTP is defined as the period elapsing between the date of randomization and the date of disease progression.
Overall survival (OS) | at randomization, then at the end of every two cycle (i.e. approximately every 8 weeks), until death from any cause. Assessed up to 24 months.
  OS is defined as the interval between time of randomization and the date of death from any cause.
Objective response rate (ORR) in each arm | At baseline, then at the end of every two cycle (i.e. approximately every 8 weeks), until disease progression or discontinuation from study. Assessed up to 24 months.
  The Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) will be used to establish disease response or progression
Disease control rate (DCR) in each arm | At baseline, then at the end of every two cycle (i.e. approximately every 8 weeks), until disease progression or discontinuation from study. Assessed up to 24 months.
  DCR will be defined as the proportion of patients achieving either partial response (PR) or complete response (CR) or stable disease (SD).
The safety and tolerability of the combination of YIV-906 plus sorafenib as measured by the rate and severity of AEs | Continuously throughout the study until 28 days after treatment discontinuation
  All patients will be evaluated and graded for adverse events according to the NCI Common Terminology for Adverse Events, version 5.0 (CTCAE).
Change of quality of life (QoL) in each arm with HCC18 | At the beginning of every course (4 weeks) until the end of study. Assessed up to 24 months.
  Each of the domains in the HCC18 will be scored per the assessment's scoring algorithm and summarized using descriptive statistics at baseline
Change of quality of life (QoL) in each arm with EORTC-C30 | At the beginning of every course (4 weeks) until the end of study. Assessed up to 24 months.
  Each of the domains in the EORTC QLQ-C30 will be scored per the assessment' scoring algorithm and summarized using descriptive statistics at baseline
Effects of YIV-906 on mean Cmax (mg/mL) of sorafenib in blood | On Day 1 of Cycle 1 (4 week/28 days), PK studied immediately prior to dose administration and at 1 hour, 2 hours, 4 hours, and 12 hours post-dose administration.
  PK is optional and limited to the first 15 male and 15 female patients from China study sites. Patients will be randomized to either study drug arm or placebo arm (2:1 ratio).
Effects of YIV-906 on mean Tmax (Hr) of sorafenib in blood | On Day 1 of Cycle 1(4 week/28 days), PK studied immediately prior to dose administration and at 1 hour, 2 hours, 4 hours, and 12 hours post-dose administration.
  PK is optional and limited to the first 15 male and 15 female patients from China study sites. Patients will be randomized to either study drug arm or placebo arm (2:1 ratio).
Effects of YIV-906 on mean AUC0-24(mg*h/L) of sorafenib in blood | On Day 1 of Cycle 1(4 week/28 days), PK studied immediately prior to dose administration and at 1 hour, 2 hours, 4 hours, and 12 hours post-dose administration.
  PK is optional and limited to the first 15 male and 15 female patients from China study sites. Patients will be randomized to either study drug arm or placebo arm (2:1 ratio).
Effects of YIV-906 on mean AUC from time 0 to the end of the dosing period AUC0-tau (mg*h/L) of sorafenib in blood | On Day 1 of Cycle 1(4 week/28 days), PK studied immediately prior to dose administration and at 1 hour, 2 hours, 4 hours, and 12 hours post-dose administration.
  PK is optional and limited to the first 15 male and 15 female patients from China study sites. Patients will be randomized to either study drug arm or placebo arm (2:1 ratio).
Effects of YIV-906 on mean t½ (Hr) of sorafenib in blood | On Day 1 of Cycle 1(4 week/28 days), PK studied immediately prior to dose administration and at 1 hour, 2 hours, 4 hours, and 12 hours post-dose administration.
  PK is optional and limited to the first 15 male and 15 female patients from China study sites.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Yen, MD/PhD, Study Chair — Taipei Medical University; Ghassan Abou-Alfa, MD/MBA, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (24):
- United States (4):
  - Calvin Pan. MD Gastroenterology & Hepatology Clinic, Flushing, New York
  - Northwell Monter Cancer Institute, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- China (12):
  - Beijing You'An Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Foshan Hospital of Traditional Chinese Medicine, Foshan, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hunan Cancer Hospital, Changsha, Hunan
  - LongHua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanghai Eastern Hepatobiliary Hospital, Shanghai, Shanghai Municipality
  - Shanghai University of Traditional Chinese Medicine Shuguang Hospital, Shanghai, Shanghai Municipality
- Queen Mary Hospital, Hong Kong, Hong Kong
- Taiwan (7):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Cancer Research Center, Taipei Municipal Wanfang Hospital, Taipei
  - Taipei Medical University -Shuang Ho Hospital, Ministry of Health and Welfare, Taipei
  - Taipei Medical University Cancer Center, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

REFERENCES:
- [Background] Lam W, Ren Y, Guan F, Jiang Z, Cheng W, Xu CH, Liu SH, Cheng YC. Mechanism Based Quality Control (MBQC) of Herbal Products: A Case Study YIV-906 (PHY906). Front Pharmacol. 2018 Nov 19;9:1324. doi: 10.3389/fphar.2018.01324. eCollection 2018. PMID 30510512
- [Background] Chu E. Wedding Rigorous Scientific Methodology and Ancient Herbal Wisdom to Benefit Cancer Patients: The Development of PHY906. Oncology (Williston Park). 2018 Feb 15;32(2):e20-e27. PMID 29492950
- [Background] Lam W, Jiang Z, Guan F, Huang X, Hu R, Wang J, Bussom S, Liu SH, Zhao H, Yen Y, Cheng YC. PHY906(KD018), an adjuvant based on a 1800-year-old Chinese medicine, enhanced the anti-tumor activity of Sorafenib by changing the tumor microenvironment. Sci Rep. 2015 Mar 30;5:9384. doi: 10.1038/srep09384. PMID 25819872
- [Background] Rockwell S, Grove TA, Liu Y, Cheng YC, Higgins SA, Booth CJ. Preclinical studies of the Chinese Herbal Medicine formulation PHY906 (KD018) as a potential adjunct to radiation therapy. Int J Radiat Biol. 2013 Jan;89(1):16-25. doi: 10.3109/09553002.2012.717733. Epub 2012 Sep 3. PMID 22856538
- [Background] Liu SH, Cheng YC. Old formula, new Rx: the journey of PHY906 as cancer adjuvant therapy. J Ethnopharmacol. 2012 Apr 10;140(3):614-23. doi: 10.1016/j.jep.2012.01.047. Epub 2012 Feb 3. PMID 22326673
- [Background] Wang E, Bussom S, Chen J, Quinn C, Bedognetti D, Lam W, Guan F, Jiang Z, Mark Y, Zhao Y, Stroncek DF, White J, Marincola FM, Cheng YC. Interaction of a traditional Chinese Medicine (PHY906) and CPT-11 on the inflammatory process in the tumor microenvironment. BMC Med Genomics. 2011 May 11;4:38. doi: 10.1186/1755-8794-4-38. PMID 21569348
- [Background] Lam W, Bussom S, Guan F, Jiang Z, Zhang W, Gullen EA, Liu SH, Cheng YC. The four-herb Chinese medicine PHY906 reduces chemotherapy-induced gastrointestinal toxicity. Sci Transl Med. 2010 Aug 18;2(45):45ra59. doi: 10.1126/scitranslmed.3001270. PMID 20720216
- [Result] Saif MW, Li J, Lamb L, Kaley K, Elligers K, Jiang Z, Bussom S, Liu SH, Cheng YC. First-in-human phase II trial of the botanical formulation PHY906 with capecitabine as second-line therapy in patients with advanced pancreatic cancer. Cancer Chemother Pharmacol. 2014 Feb;73(2):373-80. doi: 10.1007/s00280-013-2359-7. Epub 2013 Dec 3. PMID 24297682
- [Result] Kummar S, Copur MS, Rose M, Wadler S, Stephenson J, O'Rourke M, Brenckman W, Tilton R, Liu SH, Jiang Z, Su T, Cheng YC, Chu E. A phase I study of the chinese herbal medicine PHY906 as a modulator of irinotecan-based chemotherapy in patients with advanced colorectal cancer. Clin Colorectal Cancer. 2011 Jun;10(2):85-96. doi: 10.1016/j.clcc.2011.03.003. Epub 2011 Apr 22. PMID 21859559
- [Result] Saif MW, Lansigan F, Ruta S, Lamb L, Mezes M, Elligers K, Grant N, Jiang ZL, Liu SH, Cheng YC. Phase I study of the botanical formulation PHY906 with capecitabine in advanced pancreatic and other gastrointestinal malignancies. Phytomedicine. 2010 Mar;17(3-4):161-9. doi: 10.1016/j.phymed.2009.12.016. Epub 2010 Jan 22. PMID 20092990
- [Result] Yen Y, So S, Rose M, Saif MW, Chu E, Liu SH, Foo A, Jiang Z, Su T, Cheng YC. Phase I/II study of PHY906/capecitabine in advanced hepatocellular carcinoma. Anticancer Res. 2009 Oct;29(10):4083-92. PMID 19846955
- [Result] Farrell MP, Kummar S. Phase I/IIA randomized study of PHY906, a novel herbal agent, as a modulator of chemotherapy in patients with advanced colorectal cancer. Clin Colorectal Cancer. 2003 Feb;2(4):253-6. doi: 10.3816/CCC.2003.n.007. No abstract available. PMID 12620148